CLINICAL TRIAL: NCT05081531
Title: Artificial Intelligence for Locally Advanced Head Neck Cancer Treated With Multi-modality Adaptive RadioTherapy: Machine Learning-based Radiomic Prediction of Outcome and Toxicity (RadiomicART)
Brief Title: AI for Head Neck Cancer Treated With Adaptive RadioTherapy (RadiomicART)
Acronym: RadiomicArt
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2986
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adaptive Radiotherapy in Head and Neck cancer patients (Other): Patients will be treated with a total dose of 66 Gy, 60 Gy and 54 Gy on PTV1, PTV2 and PTV3, respectively, delivered in 30 fractions, 5 fractions per week.
  At week 3 from RT start, patients will repeat contrast simulation CT with, and MRI and FDG-PET scan for treatment replanning. Patient will start with the new plan in week 4.
  Interventions: Radiation: Adaptive Radiotherapy

INTERVENTIONS:
Radiation: Adaptive Radiotherapy — All the patients will be treated with VMAT technique in its RapidArc form. A simultaneous integrated boost (SIB) technique will be used. The GTV will encompass the tumor delineated on CT scan, adjusted for MRI and PET scans. Patients will be treated with a total dose of 66 Gy, 60 Gy and 54 Gy on PTV1, PTV2 and PTV3, respectively, delivered in 30 fractions, 5 fractions per week.

SUMMARY:
Current clinical management algorithms for squamous cell carcinoma of head and neck (HNSCC) involve the use of surgery and / or radiotherapy (RT) depending on the stage of the disease at diagnosis. Radical RT, exclusive or in combination with systemic therapy, represents an effective therapeutic option according to the international guidelines. Despite the recent technological advancements in the field of RT, about 30-50% of patients will develop locoregional failure after primary treatment . Moreover, although the development of Intensity modulated radiation therapy (IMRT) and Volumetric modulated arc therapy (VMAT) techniques allowed a greater sparing of dose on healthy tissues, radiation-induced toxicity still represents a relevant concern, impacting on quality of life. The continuous effort of personalized medicine has the goal of improving patient's outcome, in terms of both disease's control and pattern of toxicity. Advanced imaging modalities appear to play an essential role in the customization of the radiation treatment as shown through the use of Adaptive Radiotherapy (ART) and radiomic. With ART we mean the adaptation of tumor volumes and surrounding organs at risk (OARs) to the shrinkage and patient emaciation during RT treatment. Adaptive radiotherapy (ART) includes techniques that allow knowledge of patient-specific anatomical variations informed by Image-guided radiotherapies (IGRTs) to feedback into the plan and dose-delivery optimization during the treatment course. Radiomic is the extraction of quantitative features from medical images to characterize tumor pathology or heterogeneity. Radiomic features extracted from medical images can be used as input features to create a machine learning model able to predict survival, and to guide treatment thanks to its predictive value in view of therapy personalization.

The combination of both ART and radiomic analysis could potentially be considered a further advance in the personalization of oncological treatments, and in particular for radiation treatments. For this reason, the investigators designed the present research project with the aim to prospectively evaluate a machine learning-based radiomic approach to predict outcome and toxicity of HNSCC patients treated with ART by mean of CT, MRI and PET-scan.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the head and neck (HNSCC) is characterized by an incidence in Europe of 140.000 new cases per year, with survival rates at 5 years ranging from 25 to 65%.

Current clinical management algorithms for HNSCC patients involve the use of surgery and / or radiotherapy depending on the stage of the disease at diagnosis. Radical radiotherapy (RT), exclusive or in combination with systemic therapy, represents an effective therapeutic option according to the international guidelines.

Despite the recent technological advancements in the field of radiation therapy, about 30-50% of patients will develop locoregional failure after primary treatment of head and neck cancer. Moreover, although the development of Intensity modulated radiation therapy (IMRT) and Volumetric modulated arc therapy (VMAT) techniques allowed a greater sparing of dose on healthy tissues, radiation-induced toxicity still represents a relevant concern, impacting on quality of life of cancer patients even for long time after treatment.

The continuous effort of personalized medicine has the goal of improving patient's outcome, in terms of both disease's control and pattern of toxicity. Advanced imaging modalities appear to play an essential role in the customization of the radiation treatment as shown through the use of Adaptive Radiotherapy (ART) and radiomic.

With ART the investigators mean the adaptation of tumor volumes and surrounding organs at risk (OARs) to the shrinkage and patient emaciation during RT treatment.

The recent literature showed that tumor shrinkage can reach 70% by the end of the RT treatment, and at the same time OARs, such as parotid glands, can reduce their size by 7 to 70%. These alterations, if not taken into account, can lead to an unexpected delivery of lower dose on the tumor and higher dose of OARs compared to what planned.

Adaptive radiotherapy (ART) includes techniques that allow knowledge of patient-specific anatomical variations informed by Image-guided radiotherapies (IGRTs) to feedback into the plan and dose-delivery optimization during the treatment course. The persisting weakest link in the treatment chain for radiotherapy remains clinician-led target identification.

Compared to CT or CBCT, MRI offers superior soft-tissue definition with no associated radiation risk. MRI identifies targets larger than on CT because tumour that otherwise would have been missed is now seenah; however, most commonly, targets are reported to be smaller when delineated on MRI. The resulting smaller MRI-derived target improves the therapeutic ratio so enabling dose escalation. The availability of 'functional' MRI sequences holds promise that geometric adaptation maybe complemented by biological adaptation. Diffusion-weighted imaging (DWI) is a functional imaging technique dependent on the random motion of water molecules to generate image contrast. As tumours usually have greater cellularity than normal tissue, they demonstrate higher signal intensity, i.e., restricted diffusion on MRI. This is reflected in the low mean apparent diffusion coefficient (ADC) value. This has potential to provide both qualitative and quantitative information. Change in the ADC has been used to identify early treatment response, and to predict local recurrence. Therefore, on-board DWI could identify early non-responders who may benefit from change in treatment approach.

Radiomic is the extraction of quantitative features from medical images to characterize tumor pathology or heterogeneity. Radiomic features extracted from medical images can be used as in put features to create a machine learning model able to predict survival, and to guide treatment thanks to its predictive value in view of therapy personalization.

We previously evaluated in a retrospective study the qualitative analysis of the radiomic characteristics of head and neck tumor tissues, in order to identify a predictive signature of the biological characteristics of the tumor. The investigators stratified HNSCC patients according to the most significant radiomic features into high- and low-risk groups of relapse and survival after radio-chemotherapy.

The combination of both ART and radiomic analysis could potentially be considered a further advance in the personalization of oncological treatments, and in particular for radiation treatments. For this reason, the investigator designed the present research project with the aim to prospectively evaluate a machine learning-based radiomic approach to predict outcome and toxicity of HNSCC patients treated with ART by mean of CT, MRI and PET-scan.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance status 0 to 2
* Life expectancy > 12 months
* Histological proven squamous cell carcinoma of the pharynx, larynx or oral cavity
* Locally advanced stage disease classified as T3-T4 or N1-3
* Radical radiotherapy +/- chemotherapy indicated as the primary treatment modality
* Visible disease at the primary site on imaging performed within 4 weeks of starting treatment
* Adequate liver function
* Adequate renal function for infusion of iv. contrast for CT-scan and MRI-scan
* Adequate bone marrow function
* Written informed consent
* No previous radiation therapy on head and neck region

Exclusion Criteria:

* Inability to provide informed consent
* Presence of distant metastases
* Previous radiation therapy on head and neck region
* Pregnant or breastfeeding patients
* Prior malignancy within the last five years (except adequately treated basal cell carcinoma of the skin or in situ carcinoma of the skin or in situ carcinoma of the cervix, surgically cured, or localized prostate cancer without evidence of biochemical progression)
* Mental conditions rendering the patient incapable to understand the nature, scope, and consequences of the study
* Allergy or contraindication to contrast agents
* General contraindications to MRI
* ECOG PS >=3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Locoregional recurrence free survival | 1 year
  Locoregional recurrence free survival in head and neck cancer patients treated with adaptive radiotherapy

SECONDARY OUTCOMES:
Progression Free Survival | 1 year
  Progression Free Survival in head and neck cancer patients treated with adaptive radiotherapy
Overall Survival | 1 year
  Overall Survival in head and neck cancer patients treated with adaptive radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Clinical institute, Rozzano, Milano, Italy